CLINICAL TRIAL: NCT00713414
Title: Role of Neurotransmission and Functional CNS Networks in Spasmodic Dysphonia and Other Focal Dystonias
Brief Title: Role of Neurotransmission and Functional CNS Networks in Spasmodic Dysphonia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080181; 08-N-0181
Record Dates: First submitted 2008-07-10; First posted 2008-07-11 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-09-21

CONDITIONS: Spasmodic Dysphonia; Focal Dystonia
Keywords: Spasmodic Dysphonia; Dystonia; Basal Ganglia; PET Imaging; fMRI; Voice Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Dysphonia; Dystonic Disorders; Dystonia; Voice Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine how the brain controls speech in patients with spasmodic dysphonia, a voice disorder that involves involuntary spasms of muscles in the larynx (voice box), causing breaks in speech. Although the causes of spasmodic dysphonia are unknown, recent studies found changes in brain function in patients with the disorder that may play a role in its development.

People between 21 and 80 years of age with adductor spasmodic dysphonia may be eligible for this study. Candidates are screened with the following procedures:

Medical history and physical examination.

Nasolaryngoscopy to examine the larynx. For this test, the inside of the subject s nose is sprayed with a decongestant and a small, flexible tube called a nasolaryngoscope is passed through the nose to the back of the throat to allow examination of the larynx. The subject may be asked to talk, sing, whistle and say prolonged vowels during the procedure. The nasolaryngoscope is connected to a camera that records the movement of the vocal cords during these tasks.

Voice and speech recording to measure the type and severity of voice disorder. Subjects are asked questions about their voice disorder and their voice is recorded while they repeat sentences and sounds.

Participants undergo positron emission tomography (PET) and magnetic resonance imaging (MRI) of the brain, as follows:

PET: A catheter is placed in a vein in the subject s arm to inject a radioactive substance called a tracer that is detected by the PET scanner and provides information on brain function. [11C]flumazenil is used in one scanning session and [11C]raclopride is used in another. For the scan, the subject lies on a bed that slides in and out of the doughnut-shaped scanner, wearing a custom-molded mask to support the head and prevent it from moving during the scan. For the first scan the subject lies quietly for 60 minutes. For the second scan, the subject lies quietly for 50 minutes and is then asked to say sentences during another 50 minutes. The amount of radiation received in this study equals to a uniform whole-body exposure of 0.9 rem, which is within the dose guideline established by the NIH Radiation Safety Committee for research subjects. The guideline is an effective dose of 5 rem received per year.

MRI: This procedure uses a strong magnetic field and radio waves instead of X-rays to obtain images of the brain. The subject lies on a table that slides into the scanner, a narrow metal cylinder, wearing ear plugs to muffle loud knocking sounds that occur during the scan. Images of the brain structure are obtained while the subject lies still in the machine for 10 minutes. This is followed by functional MRI (fMRI) for 60 minutes, in which pictures are taken while the subject speaks, showing changes in brain regions that are involved in speech production.

DETAILED DESCRIPTION:
Spasmodic dysphonia (SD) and writer s cramp (WC) are primary focal dystonias with selective impairment of voluntary control of speaking and writing, respectively. Although the pathophysiology of SD and WC is unknown, dystonia is considered to be a disorder of basal ganglia that leads to secondary cortical and subcortical sensorimotor dysfunction. Results of recent neuroimaging studies have established microstructural abnormalities, as well as alterations of functional activity and neurotransmission within the basal ganglia-thalamo-cortical circuitry during symptom production in these patients. Abnormal functional relationships between these brain regions may play an important role in the pathophysiology of dystonia. However, the organization of functional networks and the neurochemical correlates underpinning their abnormalities have not, to date, been fully investigated. A few pharmacological reports of patients have provided indirect evidence of the contributing role of the major basal ganglia neurotransmitters, >=-aminobutyric acid (GABA) and dopamine, to the pathophysiology of this disorder. We identified decreased D2/D3 receptor binding at rest and abnormal dopamine release during both symptomatic and asymptomatic tasks in SD and WC compared to controls. We also identified altered GABAergic transmission, especially involving the laryngeal and hand sensorimotor cortex. These changes in neurotransmission may, in turn, be coupled with abnormalities of network functional activity in these patients and thus contribute to the pathophysiology of this disorder. There is, therefore, a critical need to further investigate the contribution of dopaminergic transmission via D1-family receptors as well as dopaminergic function of substantia nigra, pars compacta (SNc), in order to fully characterize abnormalities of dopaminergic neurotransmission in this disorder. Filling this knowledge gap is essential for development of effective neuropharmacological treatments for patients with SD and WC, which are limited, to date, to only short-term benefits from injections of botulinum toxin into the affected muscles every 3-4 months for a lifetime.

Objective

The objective of this application is to determine the role played by major basal ganglia neurotransmitters in the pathophysiology of primary focal dystonia. The central hypothesis is that dopaminergic transmission is selectively altered within the nigro-striatal and direct basal ganglia pathways and is correlated with abnormal dopaminergic function within the indirect basal ganglia circuitry in SD and WC patients.

Study Population:

We plan to examine patients with adductor SD (ADSD) compared to two other groups of subjects: (1) patients with another form of task-specific focal dystonia (writer s cramp, WC) and (2) healthy volunteers without history of neurological, psychiatric, or head and neck disorders. The research volunteers may be spouses of persons with SD and WC without a familial relationship.

Design:

This is a natural history study. Using neuroimaging techniques (positron emission tomography (PET), the central hypothesis will be tested by pursuing two specific aims: (1) to map the D1-like dopaminergic receptor binding in SD and WC patients as measured with PET using [11C]NNC-112; (2) to map the nigro-strital dopaminergic function in SD and WC patients as measured with PET using [18F]FDOPA.

Outcome Measures:

These studies will determine neurotransmitter function in patients with ADSD and WC compared to healthy subjects. The proposed research is expected to advance our understanding of the pathophysiology of voluntary motor control of voice and hand movements in diseased individuals as an important step in identifying possible mechanisms for potential neuropharmacological interventions in these patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy research volunteers and adult patients with ADSD and WC will be eligible for the study.

1. Adult patients with ADSD will have clinically documented ADSD established by voice and speech testing and fiberoptic nasolaryngoscopy.

   Patients will be required to have:
   * Intermittent uncontrolled voice breaks in vowels, liquids (r & l), semivowels (w & y) during speech in ADSD (at least 3 voice breaks), or
   * Less prominent symptoms during whisper, singing, falsetto, or shout;
   * Normal voice and vocal fold movement during protective laryngeal functions and emotional phonation, such as cough, laughter, cry.
2. Adult patients with WC will have clinically documented WC established by history and neurological examination.
3. Controls will be healthy subjects with a negative history of laryngeal, neurological, or psychiatric problems.
4. All participants will be from 21 to 80 years old and right hand dominant.
5. All participants should be able to perform a sequential finger-tapping task for 40 seconds consecutively

EXCLUSION CRITERIA:

1. Subjects who are incapable of giving an informed consent.
2. Pregnant or breastfeeding women until a time when they are no longer pregnant or breastfeeding.
3. Subjects with past or present medical history of (a) neurological problems, such as stroke, movement disorders (other than SD and WC in the patient group), brain tumors, traumatic brain injury with loss of consciousness, ataxias, myopathies, myasthenia gravis, demyelinating diseases, alcoholism, drug dependence; (b) psychiatric problems, such as schizophrenia, major and/or bipolar depression, obsessive-compulsive disorder; (c) laryngeal problems, such as vocal fold paralysis, paresis, vocal fold nodules and polyps, carcinoma, chronic laryngitis. (d) ventricular arrhythmias, renal and hepatic insufficiency, vascular headache, or carcinoid syndrome.
4. Patients who are currently taking medications known to affect GABA and dopamine receptor binding. Occasionally, patients report receiving such medication, although dopaminergic and GABA agonist/antagonists are not typically prescribed in these patients.
5. Patients who received treatment with botulinum toxin injections into the laryngeal muscles within the past 3 months.
6. Patients with vocal and hand tremor or muscle tension dysphonia.
7. Subjects who have tattoos with contraindications to MRI, ferromagnetic objects in their bodies (e.g., implanted stimulators, surgical clips, prosthesis, artificial heart valve, etc.) that cannot be removed for the purpose of study participation.
8. Subjects who received previous radiation exposure greater than 5.0 rem per year.
9. WC patients who experience focal hand dystonia at rest.
10. WC patients who have focal hand dystonia associated with trauma or a known neuroanatomic lesion or disease.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-07-09; Study Completion 2016-09-21

PRIMARY OUTCOMES:
Identify GABAergic and dopaminergic transmission in patients with spasmodic dysphonia and healthy subjects

SECONDARY OUTCOMES:
Determine the functional brain networks during speech and at rest in patients with spasmodic dysphonia compared to healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Albin RL, Young AB, Penney JB. The functional anatomy of basal ganglia disorders. Trends Neurosci. 1989 Oct;12(10):366-75. doi: 10.1016/0166-2236(89)90074-x. PMID 2479133
- [Background] Alexander GE, Crutcher MD. Functional architecture of basal ganglia circuits: neural substrates of parallel processing. Trends Neurosci. 1990 Jul;13(7):266-71. doi: 10.1016/0166-2236(90)90107-l. PMID 1695401
- [Background] Ali SO, Thomassen M, Schulz GM, Hosey LA, Varga M, Ludlow CL, Braun AR. Alterations in CNS activity induced by botulinum toxin treatment in spasmodic dysphonia: an H215O PET study. J Speech Lang Hear Res. 2006 Oct;49(5):1127-46. doi: 10.1044/1092-4388(2006/081). PMID 17077220